CLINICAL TRIAL: NCT00366041
Title: Multicentre Clinical Study to Compare the Efficacy and the Tolerance of Cellularised LG002 With the Efficacy and Tolerance of Uncellularised LG002 in the Treatment of Severe Burn Injury
Brief Title: Efficacy and Tolerance of Cellularised LG002 Versus Uncellularised LG002 in the Treatment of Severe Burns Injuries
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not appropriate to carry on the study
Sponsor: Laboratoires Genévrier (Industry)
Collaborators: Hôpital d'Instruction des Armées de Percy (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Laboratoires Genévrier, sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 03F/DE01
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cellularised LG002 (Experimental): Cellularised LG002
  Interventions: Drug: Dermal substrate cellularised LG002 (10x10cm)
- UnCellularised LG002 (Experimental): UnCellularised LG002
  Interventions: Device: Dermal substrate uncellularised LG002 (10x10 cm)

INTERVENTIONS:
Drug: Dermal substrate cellularised LG002 (10x10cm) — application depending on burn injury surface
  Arms: Cellularised LG002
Device: Dermal substrate uncellularised LG002 (10x10 cm) — depending on burn injury surface
  Arms: UnCellularised LG002

SUMMARY:
After severe burn injury, the full-thickness burn areas are excised (in the first week) and then temporarily covered with allograft (cryogenic preserved cadaver skin). This first covering is then replaced with thin skin meshed autograft.

In this study, either the dermal substrates cellularised LG002 or uncellularised LG002 will be grafted, after excision, in symmetrical areas, in replacement of the allografts. Fourteen to twenty one days after this first covering, the dermal substrate will be covered with thin skin meshed autograft.

DETAILED DESCRIPTION:
For lesions that cannot heal spontaneously, the wound is excised until fascia. Four contiguous dermal substrates (uncellularised and cellularised) are randomly grafted on each symmetric area.

A primary siliconized dressing will cover the wound. Secondary dressing: dressing gauze impregnated with physiologic serum and/or sterile dried dressing gauze, the whole is maintained by a (slightly compressive) tubular or elastic bandage.

Thin skin meshed autograft will occur 14 to 21 days after dermal substrate cellularised LG002 or uncellularised LG002 grafting (time frame necessary for the site to vascularize).

Meshed autograft development must be identical in both symmetric areas, for one single patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe burn injuries ≥ 40 % of TBSA (Total Body Surface Area)
* Thermal burn on symmetrical areas allowing grafting of 4 contiguous dermal substrates (cellularised LG002 or uncellularised LG002) on each area
* The patient himself, or his legal representative, must give his informed consent in writing

Exclusion Criteria:

* Anterior progressive serious illness (i.e severe hepatic insufficiency, immunodepression induced by corticotherapy or illness (AIDS))
* Metabolic disease
* Systemic infection or local burn infection
* Known allergy to collagen, streptomycin, Penicillin and/or bovine origine products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of take of thin skin autografts 6 days after their application on dermal substrate cellularised LG002 or uncellularised LG002 (visual assessment + photography) | 6 days after their application on dermal substrate cellularised LG002 or uncellularised LG002

SECONDARY OUTCOMES:
Short and medium term: Percentage of take of thin skin autografts 12 and 30 days after their application | 12 and 30 days after their application
Long term: Clinical evaluation (Vancouver scale 1, 3, 6, 12 months) and histological evaluation (3mm biopsy) to investigate the dermal-epidermal junction and the extra-cellular matrix (1 and 6 month) in order to evaluate the scar quality | 1, 3, 6, 12 months
Tolerance parameter: Investigator's global judgement, post grafting infection (swabbing during each new dressing for staphylococcus aureus detection), adverse event for intolerance | each application
Supplementary parameter: Allogenic fibroblasts survival : chimerism study with biopsy (1 and 6 months) | 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine DOSQUET, MD, Study Chair — Hôpital Saint Louis, Unité thérapie cellulaire et Unité INSERM 553; Daniel WASSERMANN, PhD, MD, Principal Investigator — Hôpital Cochin, Service des Brûlés
Locations (2):
- France (2):
  - Hôpital d' Instruction des Armées de Percy, Service des Brûlés, Clamart
  - Hôpital Cochin, Service des Brûlés, Paris

REFERENCES:
- [Background] Berthod F, Saintigny G, Chretien F, Hayek D, Collombel C, Damour O. Optimization of thickness, pore size and mechanical properties of a biomaterial designed for deep burn coverage. Clin Mater. 1994;15(4):259-65. doi: 10.1016/0267-6605(94)90055-8. PMID 10147169
- [Background] Damour O, Gueugniaud PY, Berthin-Maghit M, Rousselle P, Berthod F, Sahuc F, Collombel C. A dermal substrate made of collagen--GAG--chitosan for deep burn coverage: first clinical uses. Clin Mater. 1994;15(4):273-6. doi: 10.1016/0267-6605(94)90057-4. PMID 10147171
- [Background] Coulomb B, Lebreton C, Dubertret L. Influence of human dermal fibroblasts on epidermalization. J Invest Dermatol. 1989 Jan;92(1):122-5. doi: 10.1111/1523-1747.ep13071335. PMID 2909624
- [Background] Berthod F, Hayek D, Damour O, Collombel C. Collagen synthesis by fibroblasts cultured within a collagen sponge. Biomaterials. 1993 Aug;14(10):749-54. doi: 10.1016/0142-9612(93)90039-5. PMID 8218724
- [Background] Froget S, Barthelemy E, Guillot F, Soler C, Coudert MC, Benbunan M, Dosquet C. Wound healing mediator production by human dermal fibroblasts grown within a collagen-GAG matrix for skin repair in humans. Eur Cytokine Netw. 2003 Jan-Mar;14(1):60-4. PMID 12799215
- [Background] Saintigny G, Bonnard M, Damour O, Collombel C. Reconstruction of epidermis on a chitosan cross-linked collagen-GAG lattice: effect of fibroblasts. Acta Derm Venereol. 1993 Jun;73(3):175-80. doi: 10.2340/0001555573175180. PMID 8105612
- [Background] Sher SE, Hull BE, Rosen S, Church D, Friedman L, Bell E. Acceptance of allogeneic fibroblasts in skin equivalent transplants. Transplantation. 1983 Nov;36(5):552-7. doi: 10.1097/00007890-198311000-00015. PMID 6356519
- [Background] Braye FM, Stefani A, Venet E, Pieptu D, Tissot E, Damour O. Grafting of large pieces of human reconstructed skin in a porcine model. Br J Plast Surg. 2001 Sep;54(6):532-8. doi: 10.1054/bjps.2001.3620. PMID 11513518
- [Background] Coulomb B, Friteau L, Baruch J, Guilbaud J, Chretien-Marquet B, Glicenstein J, Lebreton-Decoster C, Bell E, Dubertret L. Advantage of the presence of living dermal fibroblasts within in vitro reconstructed skin for grafting in humans. Plast Reconstr Surg. 1998 Jun;101(7):1891-903. doi: 10.1097/00006534-199806000-00018. PMID 9623833